CLINICAL TRIAL: NCT05630040
Title: Vagus Nerve Simulation for Long-COVID-19
Brief Title: VNS for Long-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Director of Rehabilitation Innovation, Mount Sinai Health System Associate Professor of Rehabilitation and Human Performance, Icahn School of Medicine at Mount Sinai, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-22-00985
Record Dates: First submitted 2022-11-21; First posted 2022-11-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Post-COVID-19 Syndrome; Postural Tachycardia Syndrome; Dysautonomia
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This will be a placebo controlled, double blind, randomized control trial with a crossover design built in.
  Those randomized to the sham group will be given the opportunity to "crossover" into the active VNS arm once they have completed the sham arm (Week 12).
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will have a blinded assessor and all participants will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non-invasive Vagus Nerve Stimulation (Experimental): Participants in the Non-Invasive Vagus Nerve Stimulation arm will have devices calibrated to a therapeutic setting.
  Interventions: Device: Non-invasive vagus nerve stimulation
- Sham Vagus Nerve Stimulation (Sham Comparator): Participants in the "sham VNS" arm will be asked to use the VNS device daily on a sham setting for six weeks and will be given the opportunity to "crossover" into the active VNS arm once they have completed the sham arm.
  Interventions: Device: Non-invasive vagus nerve stimulation; Device: Sham Intervention

INTERVENTIONS:
Device: Non-invasive vagus nerve stimulation — Participants will take the VNS device home and asked to perform a daily VNS protocol designed to down regulate sympathetic nervous system activity for 6 weeks.
  Other Names: Vagus nerve stimulation
Device: Sham Intervention — Participants will take a placebo device home for 6 weeks and use daily.
  Arms: Sham Vagus Nerve Stimulation

SUMMARY:
The goal of this proposed clinical case series is to evaluate the effect of a non-invasive vagus nerve stimulation paradigm on: 1) Symptom reporting via validated patient reported outcomes, and 2) objective clinical biomarkers of autonomic nervous system function.

This will be a placebo controlled, randomized controlled trial with a crossover design built in. This study will aim to recruit 40 people with Long COVID to be a part of this research.

DETAILED DESCRIPTION:
Participants will be randomized into one of two arms. Those in the "active VNS" arm will be sent home with a portable VNS device and asked to perform a daily VNS protocol designed to down regulate sympathetic nervous system activity for six weeks.

Those in the "sham VNS" arm will be asked to use the VNS device daily on a sham setting for six weeks. Those randomized to the sham group will be given the opportunity to "crossover" into the active VNS arm once they have completed the sham arm (Week 12). The participant and assessor will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* At least 18 years of age
* Clinical diagnosis of dysautonomia following an acute COVID-19 infection at least 3 months prior. See below for criteria:

  * clinical diagnosis of autonomic dysfunction as evaluated by a qualified healthcare provider
* 2 or more if the following clinical assessment findings
* symptomatic exacerbation during active stand test
* tachycardia on active stand test
* tachycardia on orthostatic vitals assessment
* hypotension on orthostatic vitals assessment
* hypertension in orthostatic vitals assessment
* symptom exacerbation on orthostatic vitals assessment
* English speaking

Exclusion Criteria:

• Pregnancy or lactation:

* Pregnant persons will not be included in this study for the following reasons:

  * There is not sufficient data surrounding the hormone cycle changes during pregnancy and its effects on the condition being studied (PCD). The results could be skewed due to pregnancy.
  * Of note, there are no risks for pregnant persons to participate.

According to the device manufacturer, the following contraindications will be followed during the screening process:

* Patients with an active implantable medical device, such as a cardiac pacemaker, heading aid implant, or any implanted metallic or electronic device
* Patients with a history of baseline cardiac disease or atherosclerotic cardiovascular disease, including congestive heath failure (CHF), known severe coronary artery disease or recent myocardial infarction (within 5 years)
* Patients with diagnosed bradycardia
* Patients who have had surgery to cut the vagus nerve in the neck (cervical vagotomy) Patients diagnosed with narrowing of the arteries (carotid atherosclerosis)
* Patients whose pain syndromes are undiagnosed
* Pediatric patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Composite Dysautonomia Symptom Score (COMPASS 31) | Baseline (Week 0)
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains.
  The total score will be between 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.
Composite Dysautonomia Symptom Score (COMPASS 31) | Week 2
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains.
  The total score will be between 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.
Composite Dysautonomia Symptom Score (COMPASS 31) | Week 5
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains.
  The total score will be between 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.
Composite Dysautonomia Symptom Score (COMPASS 31) | Week 8
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains.
  The total score will be between 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.
Composite Dysautonomia Symptom Score (COMPASS 31) | Week 12
  COMPASS-31 (the composite autonomic symptom) score is a self-rating questionnaire evaluating six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains.
  The total score will be between 0 to 100, and a higher score indicates more severe autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, is internally consistent and applies a much-simplified scoring algorithm suitable for widespread use in autonomic research and practice.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline (Week 0)
  The Fatigue Severity Scale measures fatigue severity. The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue.
Fatigue Severity Scale (FSS) | Week 2
  The Fatigue Severity Scale measures fatigue severity. The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue.
Fatigue Severity Scale (FSS) | Week 5
  The Fatigue Severity Scale measures fatigue severity. The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue.
Fatigue Severity Scale (FSS) | Week 8
  The Fatigue Severity Scale measures fatigue severity. The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue.
Fatigue Severity Scale (FSS) | Week 12
  The Fatigue Severity Scale measures fatigue severity. The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue.
Neuro Quality of Life Score | Baseline (Week 0)
  The NeuroQOL is a self-report of health-related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five-option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Neuro Quality of Life Score | Week 2
  The NeuroQOL is a self-report of health-related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five-option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Neuro Quality of Life Score | Week 5
  The NeuroQOL is a self-report of health-related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five-option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Neuro Quality of Life Score | Week 8
  The NeuroQOL is a self-report of health-related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five-option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Neuro Quality of Life Score | Week 12
  The NeuroQOL is a self-report of health-related quality of life in 17 domains and sub-domains for adults. Item banks consist of 302 items in total (range from 5 to 45) which are used adaptively to test a variable number and content of items in a computer assisted testing format. All items are rated on a five-option scale based on intensity (e.g. 1 = not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much) or frequency ("never" to "always"). Raw scores are converted based on consistent metric (T-distribution) with data from the US general population with a T-score mean of 50 and standard deviation of 10.
Medical Research Council (MRC) Dyspnoea Scale | Baseline (Week 0)
  The MRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). Full scale from 1-5, with higher score indicating more severe symptoms.
Medical Research Council (MRC) Dyspnoea Scale | Week 2
  The MRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). Full scale from 1-5, with higher score indicating more severe symptoms.
Medical Research Council (MRC) Dyspnoea Scale | Week 5
  The MRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). Full scale from 1-5, with higher score indicating more severe symptoms.
Medical Research Council (MRC) Dyspnoea Scale | Week 8
  The MRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). Full scale from 1-5, with higher score indicating more severe symptoms.
Medical Research Council (MRC) Dyspnoea Scale | Week 12
  The MRC breathlessness scale comprises ﬁve statements that describe almost the entire range of respiratory disability from none (Grade 1) to almost complete incapacity (Grade 5). Full scale from 1-5, with higher score indicating more severe symptoms.
Post-Exertional Malaise (PEM) Screener | Baseline (Week 0)
  Post-exertional malaise (PEM) is the worsening of symptoms following even minor physical or mental exertion, with symptoms typically worsening 12 to 48 hours after activity and lasting for days or even weeks. The PEM assesses symptom frequency and severity over a 6-month look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. Total score ranges 0-40, with higher scores indicate worse health outcomes.
Post-Exertional Malaise (PEM) Screener | Week 2
  Post-exertional malaise (PEM) is the worsening of symptoms following even minor physical or mental exertion, with symptoms typically worsening 12 to 48 hours after activity and lasting for days or even weeks. The PEM assesses symptom frequency and severity over a 6-month look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. Higher scores indicate worse health outcomes. Total score ranges 0-40, with higher scores indicate worse health outcomes.
Post-Exertional Malaise (PEM) Screener | Week 5
  Post-exertional malaise (PEM) is the worsening of symptoms following even minor physical or mental exertion, with symptoms typically worsening 12 to 48 hours after activity and lasting for days or even weeks. The PEM assesses symptom frequency and severity over a 6-month look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. Higher scores indicate worse health outcomes. Total score ranges 0-40, with higher scores indicate worse health outcomes.
Post-Exertional Malaise (PEM) Screener | Week 8
  Post-exertional malaise (PEM) is the worsening of symptoms following even minor physical or mental exertion, with symptoms typically worsening 12 to 48 hours after activity and lasting for days or even weeks. The PEM assesses symptom frequency and severity over a 6-month look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. Higher scores indicate worse health outcomes. Total score ranges 0-40, with higher scores indicate worse health outcomes.
Post-Exertional Malaise (PEM) Screener | Week 12
  Post-exertional malaise (PEM) is the worsening of symptoms following even minor physical or mental exertion, with symptoms typically worsening 12 to 48 hours after activity and lasting for days or even weeks. The PEM assesses symptom frequency and severity over a 6-month look back period. Frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time. Severity is also rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. Total score ranges 0-40, with higher scores indicate worse health outcomes.
EQ-5D-5L Quality of Life Score | Baseline (Week 0)
  The EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state, thus, higher scores indicate better health outcomes.
EQ-5D-5L Quality of Life Score | Week 2
  The EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state, thus, higher scores indicate better health outcomes.
EQ-5D-5L Quality of Life Score | Week 5
  The EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state, thus, higher scores indicate better health outcomes.
EQ-5D-5L Quality of Life Score | Week 8
  The EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state, thus, higher scores indicate better health outcomes.
EQ-5D-5L Quality of Life Score | Week 12
  The EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state, thus, higher scores indicate better health outcomes.
Plasma IL-6 levels | Baseline (Week 0)
  Plasma IL-6 levels as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-6 levels | Week 2
  Plasma IL-6 levels as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body in different ways.
Plasma IL-6 levels | Week 5
  Plasma IL-6 levels as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-6 levels | Week 8
  Plasma IL-6 levels as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-6 levels | Week 12
  Plasma IL-6 levels as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-1 levels | Baseline (Week 0)
  Plasma IL-1 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-1 levels | Week 2
  Plasma IL-1 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-1 levels | Week 5
  Plasma IL-1 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-1 levels | Week 8
  Plasma IL-1 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-1 levels | Week 12
  Plasma IL-1 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-10 levels | Baseline (Week 0)
  Plasma IL-10 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-10 levels | Week 2
  Plasma IL-10 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-10 levels | Week 5
  Plasma IL-10 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-10 levels | Week 8
  Plasma IL-10 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma IL-10 levels | Week 12
  Plasma IL-10 levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma HS-CRP levels | Baseline (Week 0)
  Plasma HS-CRP levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma HS-CRP levels | Week 2
  Plasma HS-CRP levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma HS-CRP levels | Week 5
  Plasma HS-CRP levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma HS-CRP levels | Week 8
  Plasma HS-CRP levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Plasma HS-CRP levels | Week 12
  Plasma HS-CRP levels: as a metric of sympathetic nervous system activation. Plasma testing evaluates for evidence of inflammation in the body.
Morning salivary cortisol levels | Baseline (Week 0)
  Morning salivary cortisol levels: As a metric of sympathetic nervous system activation. Morning salivary cortisol levels evaluate changes in the body's waking hormone responses, which indicate changes in nervous system activation in response to the intervention.
Morning salivary cortisol levels | Week 2
  Morning salivary cortisol levels: As a metric of sympathetic nervous system activation. Morning salivary cortisol levels evaluate changes in the body's waking hormone responses, which indicate changes in nervous system activation in response to the intervention.
Morning salivary cortisol levels | Week 5
  Morning salivary cortisol levels: As a metric of sympathetic nervous system activation. Morning salivary cortisol levels evaluate changes in the body's waking hormone responses, which indicate changes in nervous system activation in response to the intervention.
Morning salivary cortisol levels | Week 8
  Morning salivary cortisol levels: As a metric of sympathetic nervous system activation. Morning salivary cortisol levels evaluate changes in the body's waking hormone responses, which indicate changes in nervous system activation in response to the intervention.
Morning salivary cortisol levels | Week 12
  Morning salivary cortisol levels: As a metric of sympathetic nervous system activation. Morning salivary cortisol levels evaluate changes in the body's waking hormone responses, which indicate changes in nervous system activation in response to the intervention.
End-tidal CO2 levels | Baseline (Week 0)
  End-tidal CO2 levels: As a metric of sympathetic nervous system activation measured using a capnograph. Patients with post-COVID dysautonomia will be hypocapnic (low end-tidal CO2). High or low levels of end-tidal CO2 can drive symptoms in patients.
End-tidal CO2 levels | Week 2
  End-tidal CO2 levels: As a metric of sympathetic nervous system activation measured using a capnograph. Patients with post-COVID dysautonomia will be hypocapnic (low end-tidal CO2). High or low levels of end-tidal CO2 can drive symptoms in patients.
End-tidal CO2 levels | Week 5
  End-tidal CO2 levels: As a metric of sympathetic nervous system activation measured using a capnograph. Patients with post-COVID dysautonomia will be hypocapnic (low end-tidal CO2). High or low levels of end-tidal CO2 can drive symptoms in patients.
End-tidal CO2 levels | Week 8
  End-tidal CO2 levels: As a metric of sympathetic nervous system activation measured using a capnograph. Patients with post-COVID dysautonomia will be hypocapnic (low end-tidal CO2). High or low levels of end-tidal CO2 can drive symptoms in patients.
End-tidal CO2 levels | Week 12
  End-tidal CO2 levels: As a metric of sympathetic nervous system activation measured using a capnograph. Patients with post-COVID dysautonomia will be hypocapnic (low end-tidal CO2). High or low levels of end-tidal CO2 can drive symptoms in patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Abilities Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

DOCUMENTS (1):
  • Informed Consent Form (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT05630040/ICF_000.pdf